CLINICAL TRIAL: NCT03346291
Title: Examining Persistence in Smokers With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Marc L. Steinberg, Ph.D., Associate Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20150001885; R21DA041163-01 (NIH)
Record Dates: First submitted 2017-11-03; First posted 2017-11-17 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Smoking Cessation; Schizophrenia; Schizo Affective Disorder
MeSH Terms: conditions — Smoking Cessation; Schizophrenia; Psychotic Disorders | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Persistence Targeted Smoking Cessation (Experimental): 8 weekly counseling sessions + 10 weeks of over-the-counter nicotine patch
  Interventions: Behavioral: counseling

INTERVENTIONS:
Behavioral: counseling — individual, weekly, smoking cessation counseling + over-the-counter nicotine patch

SUMMARY:
All participants will receive free weekly counseling (8- weeks) and free nicotine patches (10-weeks). They will complete assessment measures commonly used in smoking cessation studies. We hope to show that this treatment is feasible in this small pilot study before comparing it to a more established treatment in a future randomized clinical trial.

DETAILED DESCRIPTION:
This study is a non-randomized trial of a new psychosocial treatment for smoking cessation (for smokers with schizophrenia) that is based on cognitive behavioral therapy for smoking cessation - a commonly used approach. Participants will receive free weekly counseling (8- weeks) and free nicotine patches (10-weeks). They will complete assessment measures commonly used in smoking cessation studies. We hope to show that this treatment is feasible in this small pilot study before comparing it to a more established treatment in a future randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 18 - 64 years old
* Must indicate commitment to quitting smoking in the next 30 days
* Must smoke at least 5 cigarettes per day for past 6-months
* Expired breath carbon monoxide (CO) > 5 to ensure daily cigarette use
* Must score < 8 (or <7 for women) on the Alcohol Use Disorders Identification Test
* Must score less than 3 on the 6-month Drug Abuse Screening Test-10
* Must provide a negative urine drug screen for cannabis, cocaine, opiates, or
* methamphetamine (Note: Participants with a positive screen for opiates may
* participate with proof of prescription for opiates.)
* Must have a diagnosis of Schizophrenia or Schizoaffective Disorder on Structured Clinical Interview
* Psychiatric illness must be stable, as indicated by no hospitalizations in previous 8 weeks, and a stable psychotropic medication regimen including a stable antipsychotic dose for 8 weeks

Exclusion Criteria:

* Must not be currently receiving tobacco dependence treatment counseling
* Must not currently be taking varenicline (Chantix)
* Must not be taking bupropion (Zyban/Wellbutrin) to quit smoking
* Must not be taking any nicotine preparations (gum, lozenge, patch, spray, inhaler) daily over the last 10 days.
* Must not report unstable angina pectoris, myocardial infarction, or significant cardiac arrhythmia (including atrial fibrillation) in the past 90 days
* Must not be pregnant, breastfeeding, or planning on becoming pregnant in the next 4-months. Women who can become pregnant may be included if using effective birth control
* Must not have pending legal matters with potential to result in jail time
* Must not be planning on moving outside local area in next 3-months

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-06-13 (Actual); Study Completion 2018-06-13 (Actual)

PRIMARY OUTCOMES:
Task Persistence - Mirror Tracing | Through end-of-treatment - approximately 8 weeks after baseline
  Number of seconds persisting on a computerized mirror tracing task (Higher number of seconds = greater persistence)
Task Persistence - Sustained Divided Attention Task | Through end-of-treatment - approximately 8 weeks after baseline
  Seconds persisting on Sustained Divided Attention Task (Higher number of seconds = greater persistence)
Task Persistence - Breath-holding | Through end-of-treatment - approximately 8 weeks after baseline
  Number of seconds persisting on a breath-holding endurance task (Higher number of seconds = greater persistence)
Task Persistence -Temperament and Character Inventory-Persistence Scale (TCI-P) | Through end-of-treatment - approximately 8 weeks after baseline
  Score on Temperament and Character Inventory-Persistence Scale (TCI-P) (Higher score = greater persistence)
Task Persistence - 2-item Task Persistence Measure | Through end-of-treatment - approximately 8 weeks after baseline
  Score on 2-item Task Persistence Measure (Higher score = greater persistence)
Task Persistence - Distress Tolerance Scale (DTS) | Through end-of-treatment - approximately 8 weeks after baseline
  Score on Distress Tolerance Scale (DTS) (Higher score = greater persistence)
Task Persistence - Thoughts About Smoking Questionnaire | Through end-of-treatment - approximately 8 weeks after baseline
  Score on the Thoughts About Smoking Questionnaire (Higher score = less persistence)
Self-reported ratings of ease of understanding and helpfulness of counseling | Through end-of-treatment - approximately 8 weeks after baseline
  percentage of participants who rate the intervention as "easy to understand" and "helpful"

CONTACTS AND LOCATIONS:
Overall Officials: Marc L Steinberg, Ph.D., Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/91/NCT03346291/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT03346291/ICF_001.pdf